CLINICAL TRIAL: NCT02550028
Title: Levetiracetam Treatment of Neonatal Seizures: A Multi-Centre Randomized Blinded Controlled Study of the Efficacy of Oral Levetiracetam as First Line Treatment for Neonatal Seizures in China
Brief Title: Levetiracetam Treatment of Neonatal Seizures
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital, Fujian of China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Maternal and Child Health Hospital of Hubei Province (Other); The Maternal & Children Health Hospital of Dehong, Yunnan of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHFudanU_NNICU3; NCT02602015 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-15 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Seizures
Keywords: Neonates; Seizure
MeSH Terms: conditions — Seizures | interventions — Levetiracetam; Phenobarbital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral levetiracetam (Experimental): Oral levetiracetam 50 mg/kg loading dose. 10 mg/kg 8 hourly maintenance
  Interventions: Drug: Oral levetiracetam
- Intravenous phenobarbital (Active Comparator): Intravenous phenobarbital 20 loading dose (add to 40 mg/kg if seizure discontrol). 5 mg/kg 24 hourly maintenance
  Interventions: Drug: Intravenous phenobarbital

INTERVENTIONS:
Drug: Oral levetiracetam — Oral load of levetiracetam (50 mg/kg) following identification of EEG confirmed neonatal seizure.
  Other Names: Keppra
  Arms: Oral levetiracetam
Drug: Intravenous phenobarbital — Intravenous load of phenobarbital (20 mg/kg)following EEG confirmation of seizure activity load.
  Other Names: phenobarbitone
  Arms: Intravenous phenobarbital

SUMMARY:
Current treatments for the brain damaging complication of neonatal seizures are unsatisfactory. A multi-centre Chinese clinical trials with the aim to using oral Levetiracetam to develop new treatment strategies for the treatment of neonatal seizures. The purpose of this study is to determine the correct oral dosing, safety and efficacy for oral Levetiracetam as first line treatment in term new born babies with seizures.

DETAILED DESCRIPTION:
This project aims to improve the treatment of neonatal seizures. Current treatments are poorly effective and have significant side effects. Levetiracetam has great potential as a treatment for neonatal seizures but is not approved for use in children less than 1 years of age by oral. This study aims to obtain essential data regarding the efficacy and safety of oral Levetiracetam in neonatal population and simultaneously to use EEG monitoring systems that facilitate seizure detection and research.

Specific aims are:

1. To determine the efficacy of oral Levetiracetam in terminating neonatal seizures by EEG in the Neonatal Neurological Intensive Care Unit (NNICU).
2. To determine dose escalation data by studying the additional efficacy of a further dose in non responders.
3. To determine additional pharmacokinetic data to confirm findings from our previous pharmacokinetic study.
4. To determine further safety data of oral Levetiracetam in neonates.

ELIGIBILITY:
Inclusion Criteria:

Neonatal seizure occurred and was proved by EEG according to abnormal discharge of brain. one or more of the following :

1. Male or female term baby with gestational >37 weeks and postnatal age < or= 28 days
2. Birthweight >2500g
3. Written informed consent of parent or guardian

Exclusion Criteria:

1. Babies who have been close to death
2. Seizure occurred by metabolic factors (hypoglycemia, hypocalcemia, electrolyte disorder)
3. Babies who have received phenobarbitone or any other anticonvulsive medication before hospitalization
4. Abnormal renal function

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
EEG | At Day 28
  Efficacy of levetiracetam by assessment of the change from baseline in EEG on Day 15.

SECONDARY OUTCOMES:
Brain Parenchyma Alterations(MRI) | At Day 28
  Efficacy of levetiracetam by assessment of the change of brain from baseline in MRI on Day 28.
Neurodevelopment(Bayley Scores) | At Day 28
  Efficacy of levetiracetam by assessment of the change from baseline to Day 28 in neurodevelopment via Bayley Scores of Infant Development Mental Development Index (BSID).
Seizure Control Days | From Day 1 to Day 28 post-dose in each period
  Efficacy of levetiracetam by assessment of seizure control days.
Number of Adverse Events（Abnormal Appearance） | From Day 1 to Day 28 post-dose in each period
  This is a composition of general appearance, abdomen, skin, head and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of Adverse Events（Abnormal Blood Pressure） | From Day 1 to Day 28 post-dose in each period
Number of Adverse Events(Pulse) | From Day 1 to Day 28 post-dose in each period
Number of Adverse Events(Respiratory) | From Day 1 to Day 28 post-dose in each period
Number of Abnormal Clinical Chemistry | From Day 1 to Day 28 post-dose in each period
  Safety of levetiracetam by assessment of safety laboratory tests.
Number of Abnormal Hematology | From Day 1 to Day 28 post-dose in each period
  Safety of levetiracetam by assessment of safety laboratory tests.
Number of Abnormal Clinical Urinalysis | From Day 1 to Day 28 post-dose in each period
  Safety of levetiracetam by assessment of safety laboratory tests.

OTHER OUTCOMES:
Rate and extent of absorption by assessment of tmax | At Day 1 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
  Comparison of tmax (time to reach maximum plasma concentration) of levetiracetam on Day 1 of each treatment period; up to 6 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose).
Rate and extent of absorption by assessment of Cmax | At Day 1 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
  Comparison of Cmax (maximum observed plasma concentration) of levetiracetam on Day 1 of each treatment period; up to 6 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose).
Rate and extent of absorption by assessment of AUC(0-4) | At Day 1 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose)
  Comparison of AUC(0-4) (Area under the plasma concentration-time curve from time zero to 4 hours after administration) of levetiracetam on Day 1 of each treatment period; up to 6 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, and 4 h post-dose).
Rate and extent of absorption by assessment of Cmax,ss of levetiracetam | At Day 14 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
  Comparison of Cmax,ss (observed maximum plasma concentration at steady state) of levetiracetam on Day 14 of each treatment period; up to 10 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose).
Rate and extent of absorption by assessment of AUC(0-24) of levetiracetam | At Day 14 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
  Comparison of AUC(0-24) (Area under the plasma concentration-time curve from time zero to 24 hours after administration) of levetiracetam on Day 14 of each treatment period; up to 10 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose).
Rate and extent of absorption by assessment of tmax,ss of levetiracetam | At Day 14 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
  Comparison of tmax,ss (time to reach maximum plasma concentration at steady state) of levetiracetam on Day 14 of each treatment period; up to 10 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose).
Rate and extent of absorption by assessment of Cavg,ss of levetiracetam | At Day 14 in each period (in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
  Comparison of Cavg,ss (average plasma concentration during a dosing interval at steady state) of levetiracetam on Day 14 of each treatment period; up to 10 samples will be collected in each period (i.e. in subjects with intensive pharmacokinetic assessments, at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose).
Rate and extent of absorption by assessment of AUC(0-last) of levetiracetam | At Day 1 and Day 14 in each period (in subjects with intensive pharmacokinetic assessments, on Day 1 at pre-dose and 15 and 30 minutes, and 1, 2 and 4 h post-dose, on Day 14 at pre-dose and 15 and 30 minutes, and 1, 2, 4, 8, 12, 16 and 24 h post-dose)
  Comparison of AUC(0-last) (Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration) of levetiracetam (i.e. in subjects with intensive pharmacokinetic assessments)
Rate and extent of absorption following multiple dose administration by assessment of Cmin of levetiracetam | At Day 1 and on Day 14 at pre-dose in each period
  Comparison of Cmin (predose concentration) of levetiracetam in each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Garrity LC, Turner M, Standridge SM. Increased levetiracetam clearance associated with a breakthrough seizure in a pregnant patient receiving once/day extended-release levetiracetam. Pharmacotherapy. 2014 Jul;34(7):e128-32. doi: 10.1002/phar.1439. Epub 2014 May 7. PMID 24807683
- [Background] Bansal S, Blalock D, Kebede T, Dean NP, Carpenter JL. Levetiracetam versus (fos)phenytoin for seizure prophylaxis in pediatric patients with intracranial hemorrhage. J Neurosurg Pediatr. 2014 Feb;13(2):209-15. doi: 10.3171/2013.10.PEDS13256. Epub 2013 Nov 29. PMID 24286154
- [Background] Fang Y, Wu X, Xu L, Tang X, Wang J, Zhu G, Hong Z. Randomized-controlled trials of levetiracetam as an adjunctive therapy in epilepsy of multiple seizure types. J Clin Neurosci. 2014 Jan;21(1):55-62. doi: 10.1016/j.jocn.2013.01.032. Epub 2013 Nov 11. PMID 24231559
- [Background] Khan O, Cipriani C, Wright C, Crisp E, Kirmani B. Role of intravenous levetiracetam for acute seizure management in preterm neonates. Pediatr Neurol. 2013 Nov;49(5):340-3. doi: 10.1016/j.pediatrneurol.2013.05.008. Epub 2013 Aug 3. PMID 23921284
- [Background] Inaba K, Menaker J, Branco BC, Gooch J, Okoye OT, Herrold J, Scalea TM, Dubose J, Demetriades D. A prospective multicenter comparison of levetiracetam versus phenytoin for early posttraumatic seizure prophylaxis. J Trauma Acute Care Surg. 2013 Mar;74(3):766-71; discussion 771-3. doi: 10.1097/TA.0b013e3182826e84. PMID 23425733
- [Background] Kanemura H, Sano F, Sugita K, Aihara M. Effects of levetiracetam on seizure frequency and neuropsychological impairments in children with refractory epilepsy with secondary bilateral synchrony. Seizure. 2013 Jan;22(1):43-7. doi: 10.1016/j.seizure.2012.10.003. Epub 2012 Nov 3. PMID 23127775
- [Background] Liu YH, Wang XL, Deng YC, Zhao G. Levetiracetam-associated aggravation of myoclonic seizure in children. Seizure. 2012 Dec;21(10):807-9. doi: 10.1016/j.seizure.2012.08.008. Epub 2012 Sep 16. PMID 22990039
- [Background] Jehi LE, Irwin AI, Kayyali H, Vadera S, Bingaman W, Najm I. Levetiracetam may favorably affect seizure outcome after temporal lobectomy. Epilepsia. 2012 Jun;53(6):979-86. doi: 10.1111/j.1528-1167.2012.03453.x. Epub 2012 Mar 29. PMID 22462729
- [Background] Steinbaugh LA, Lindsell CJ, Shutter LA, Szaflarski JP. Initial EEG predicts outcomes in a trial of levetiracetam vs. fosphenytoin for seizure prevention. Epilepsy Behav. 2012 Mar;23(3):280-4. doi: 10.1016/j.yebeh.2011.12.005. Epub 2012 Feb 16. PMID 22342434
- [Background] Auvin S, Chhun S, Berquin P, Ponchel E, Delanoe C, Chiron C. Aggravation of absence seizure related to levetiracetam. Eur J Paediatr Neurol. 2011 Nov;15(6):508-11. doi: 10.1016/j.ejpn.2011.05.007. Epub 2011 Jun 15. PMID 21680209